CLINICAL TRIAL: NCT00451893
Title: An Expertise-based Multicentre Randomized Controlled Trial Comparing a Heavy-weight and a Light-weight Mesh in the Operation of Inguinal Hernia
Brief Title: The Significance of the Mesh Thickness in the Operation of Inguinal Hernia
Acronym: LJUNO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Collaborators: Norrlandstingens Regionförbund (Other); Jämtland County Council, Sweden (Other Government); Västerbotten County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Markku Haapamaki, Associate professor, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LJUNO 05-109M
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; polypropylene mesh; heavy-weight mesh; light-weight mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heavy-weight (Active Comparator): Lichtenstein operation performed with a heavy-weight mesh.
  Interventions: Procedure: Lichtenstein operation with a heavy-weight mesh
- Light-weight (Active Comparator): Lichtenstein operation performed with a light-weight mesh.
  Interventions: Procedure: Lichtenstein operation with a light-weight mesh

INTERVENTIONS:
Procedure: Lichtenstein operation with a heavy-weight mesh — Bard flat mesh, polypropylene, 7,5 x 15 cm, 90 g/m2
  Arms: Heavy-weight
Procedure: Lichtenstein operation with a light-weight mesh — Johnson&Johnson Ultrapro, polypropylene/poliglecaprone, 10 x 15 cm, 28 g/m2
  Arms: Light-weight

SUMMARY:
The trial compares the postoperative complain, pain, quality of life after the implantation of a heavy-weight alternative light-weight mesh, by randomly allocating patients with inguinal hernia disease to two groups of surgeons, each group being trained to operate with one of the above mentioned meshes.

Hypothesis: There is less postoperative pain after the implantation of a light-weight mesh.

DETAILED DESCRIPTION:
The implantation of mesh in the operation of inguinal hernia has resulted in a continuously diminishing frequency of reoperations. Randomized controlled trials indicate that hernia repair with an open mesh technique has a shorter learning curve, is cheaper and may give less recurrences than laparoscopic hernia repair in general surgical practice. Furthermore, local anesthesia has significant advantages for both the patient and the health related economy compared to general anesthesia and regional anesthesia. The experience of the last decade within the field of groin hernia surgery has focused interest on quality of life and postoperative pain (especially chronic pain). Chronic pain is defined as pain that remains 3 months after the operation. Recent studies indicate that one third of all patients operated on for inguinal hernia have some degree of chronic pain and that 4-6 % of patients have pain interfering with daily activities one year after surgery.

In the present study a heavy-weight polypropylene mesh will be compared with a light-weight partly absorbable mesh. In an expertise-based randomized control trial patients will be randomly allocated to two groups of surgeons, each group well trained to use one of the two meshes.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 25 years or older
* Reducible, unilateral, inguinal hernia (not femoral hernia) that has not been operated on before

Exclusion Criteria:

* The patient is not able or do not want to give written informed consent
* The patient is not suitable for an operation in local anesthesia
* Anticoagulant medication or a known coagulation disorder

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life | Two, seven and eleven postoperative days. Four months and one year after the operation.
Pain | Two, seven and eleven postoperative days. Four months and one year after the operation.

SECONDARY OUTCOMES:
Postoperative complications | Four months and one year after the operation.
Recurrences | Four months and one year after the operation.
Health-care costs | Four months and one year after the operation.
Sick leave | Four months and one year after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Markku M Haapamaki, MD, PhD, Principal Investigator — Umeå University, Department of Surgical and Perioperative Sciences; Erik Nilsson, MD, Ph D, Study Director — Umeå University, Department of Surgical and Perioperative Sciences; Pär Nordin, MD, PhD, Principal Investigator — Umeå University, Department of Surgical and Perioperative Sciences; Rojda Gumuscu, MD, Principal Investigator — Umeå University, Department of Surgical and Perioperative Sciences; Martin Rutegård, MD, PhD, Principal Investigator — Umeå University, Department of Surgical and Perioperative Sciences
Locations (2):
- Sweden (2):
  - Östersund Hospital, Östersund
  - Department of Surgical and Perioperativ Sciences, Umeå University Hospital, Umeå

REFERENCES:
- [Derived] Rutegard M, Lindqvist M, Svensson J, Nordin P, Haapamaki MM. Chronic pain after open inguinal hernia repair: expertise-based randomized clinical trial of heavyweight or lightweight mesh. Br J Surg. 2021 Mar 12;108(2):138-144. doi: 10.1093/bjs/znaa049. PMID 33711123
- [Derived] Rutegard M, Gumuscu R, Stylianidis G, Nordin P, Nilsson E, Haapamaki MM. Chronic pain, discomfort, quality of life and impact on sex life after open inguinal hernia mesh repair: an expertise-based randomized clinical trial comparing lightweight and heavyweight mesh. Hernia. 2018 Jun;22(3):411-418. doi: 10.1007/s10029-018-1734-z. Epub 2018 Jan 20. PMID 29353339